CLINICAL TRIAL: NCT05452473
Title: Clinical Benefit in the CDSS-assisted Screening Upper Gastrointestinal Endoscopy vs. Routine Screening Endoscopy
Brief Title: CDSS-assisted UGI Endoscopy vs. Routine Screening Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Chang Seok Bang, PI, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AI RCT1
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Healthy Individual
Keywords: Convolutional neural network; Deep learning; Endoscopy; Gastric neoplasms
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDSS-assisted screening endoscopy (Experimental): Participants will be tested for CDSS-assisted screening upper gastrointestinal endoscopy
  Interventions: Other: CDSS-assisted upper GI endoscopy
- Conventional routine screening endoscopy (Placebo Comparator): Participants will be tested for Conventional routine screening upper gastrointestinal endoscopy
  Interventions: Other: no intervention

INTERVENTIONS:
Other: CDSS-assisted upper GI endoscopy — Expert endoscopists perform screening upper gastrointestinal endoscopy while looking at the monitor (CDSS system: automatic detection or lesion classification function) and listening to the sound of the monitor next to the original endoscopy monitor system.
  Arms: CDSS-assisted screening endoscopy
Other: no intervention — Expert endoscopists perform routine screening upper gastrointestinal endoscopy without CDSS's help.
  Arms: Conventional routine screening endoscopy

SUMMARY:
This study aimed to find the CDSS-assisted upper GI endoscopy has clinical benefit compared to conventional routine screening upper GI endoscopy. Investigators will conduct a pilot randomized controlled study. Consecutive patients will be allocated either to CDSS-assisted upper GI endoscopy or conventional routine screening upper GI endoscopy. The lesion detection rate will be compared between both groups.

DETAILED DESCRIPTION:
Artificial intelligence has been adopted in the field of gastrointestinal endoscopy. Investigators previously established deep-learning models to predict the histology and invasion depth of gastric lesions using endoscopic stillcut images. However, clinical benefit of this model has not been evaluated. This study aimed to find the CDSS-assisted upper GI endoscopy has clinical benefit compared to conventional routine screening upper GI endoscopy. Investigators will conduct a pilot randomized controlled study. Consecutive patients who visited Chuncheon Sacred Heart hospital will be allocated either to CDSS-assisted upper GI endoscopy or conventional routine screening upper GI endoscopy. The lesion detection rate will be compared between both groups. Expert endoscopists will conduct this randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who visited for routine screening upper gastrointestinal endoscopy

Exclusion Criteria:

* Participants who refuse to participate in this study
* Participants who showed paradoxical reaction prohibiting routine examination

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2022-08-06 (Estimated); Study Completion 2022-12-06 (Estimated)

PRIMARY OUTCOMES:
Gastric lesion detection rate | Baseline (gold standard; ground truth is expert endoscopists' lesion detection)
  Gastric lesions (low or high grade dysplasia, early gastric cancer, or advanced gastric cancer) detection rate

SECONDARY OUTCOMES:
Lesion classification accuracy | Baseline (gold standard; ground truth is histologic diagnosis of detected lesions)
  Whether CDSS correctly diagnosed detected lesions or not

CONTACTS AND LOCATIONS:
Overall Officials: Chang Seok Bang, MD, PhD, Principal Investigator — Hallym University
Locations (1):
- Chuncheon Sacred Heart hospital, Chuncheon, Gangwon-do, South Korea

REFERENCES:
- [Derived] Gong EJ, Bang CS, Lee JJ, Baik GH, Lim H, Jeong JH, Choi SW, Cho J, Kim DY, Lee KB, Shin SI, Sigmund D, Moon BI, Park SC, Lee SH, Bang KB, Son DS. Deep learning-based clinical decision support system for gastric neoplasms in real-time endoscopy: development and validation study. Endoscopy. 2023 Aug;55(8):701-708. doi: 10.1055/a-2031-0691. Epub 2023 Feb 8. PMID 36754065